CLINICAL TRIAL: NCT00184028
Title: Phase II Trial of Taxotere and Oxaliplatin Combination Chemotherapy in Squamous Cell Carcinoma of the Head and Neck
Brief Title: Combination of Taxotere and Oxaliplatin in Squamous Cell Carcinoma of the Head and Neck
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient Accrual
Sponsor: University of Southern California (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7H-03-1
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Results first posted 2013-05-06 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-05

CONDITIONS: Carcinoma of the Head and Neck
MeSH Terms: interventions — Docetaxel; Oxaliplatin

ARMS (1):
- Arm 1 (Experimental): On Day 1 of each day treatment cycle, patients receive Taxotere 60 mg/m2 as a 1-hour IV infusion, followed by the administration of oxaliplatin 100 mg/m2. Oxaliplatin will be administered IV over 2 hours at a rate of 10mg/m2/min. This treatment regimen will be repeated every 21 days.
  Interventions: Drug: Taxotere; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Taxotere — Taxotere is given at 60 mg/m2 as a 1-hour intravenous infusion.
Drug: Oxaliplatin — Oxaliplatin will be administered intravenously over 2 hours at a rate of 10mg/m2/min. on day 1 every 3 weeks.

SUMMARY:
This research study is for subjects with squamous cell cancer of the head and neck which is not solely treatable with surgery or radiation. This research study involves treatment with an experimental chemotherapy combination of oxaliplatin and Taxotere. Tha main purpose of this study is to assess the effectiveness of this combination of medications for this type of cancer.

Approximately 54 subjects will take part in this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed Head and Neck Squamous Cell Carcinoma which is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective.
* Tissue from tumor must be available. This may be paraffin embedded tissue from previous biopsy/resection. If it is not available, a repeat biopsy must be performed.
* Age greater than or equal to 18 years
* ECOG performance status less than or equal to 2 (Karnofsky greater than or equal to 50%)
* Patients must have adequate organ and marrow function as defined below:
* leukocytes greater than or equal to 3,000/microliter
* hemoglobin greater than or equal to 8.0 g/dl
* absolute neutrophil count greater than or equal to 1,500/microliter
* platelets greater than or equal to 100,000/microliter
* total bilirubin within normal institutional limits
* creatinine within normal institutional limits OR creatinine clearance greater than or equal to 60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
* If:

  * ALK PHOS is less than or equal to ULN and AST or ALT is less than or equal to ULN, patient is eligible.
  * ALK PHOS is less than or equal to ULN and AST or ALT is greater than 1x but less than or equal to 1.5x, patient is eligible.
  * ALK PHOS is less than or equal to ULN and AST or ALT is greater than 1.5x but less than or equal to 5x, patient is eligible.
  * ALK PHOS is less than or equal to ULN and AST or ALT is greater than 5x ULN, patient is ineligible.
  * ALK PHOS is greater than 1x but less than or equal to 2.5x and AST or ALT is less than or equal to ULN, patient is eligible.
  * ALK PHOS is greater than 1x but less than or equal to 2.5x and AST or ALT is greater than 1x but less than or equal to 1.5x, patient is eligible.
  * ALK PHOS is greater than 1x but less than or equal to 2.5x and AST or ALT is greater than 1.5x but less than or equal to 5x, patient is ineligible.
  * ALK PHOS is greater than 1x but less than or equal to 2.5x and AST or ALT is greater than 5x ULN, patient is ineligible.
  * ALK PHOS is greater than 2.5x but less than or equal to 5x and ALT or AST is less than or equal to ULN,patient is eligible.
  * ALK PHOS is greater than 2.5x but less than or equal to 5x and ALT or AST is greater than 1x but less than or equal to 1.5x, patient is ineligible.
  * ALK PHOS is greater than 2.5x but less than or equal to 5x and ALT or AST is greater than 1.5x but less than or equal to 5x, patient is ineligible.
  * ALK PHOS is greater than 2.5x but less than or equal to 5x and ALT or AST is greater than 5x ULN, patient is ineligible.
  * ALK PHOS is greater than 5x ULN and AST or ALT is less than or equal to ULN, patient is ineligible.
  * ALK PHOS is greater than 5x ULN and AST or ALT is greater than 1x but less than or equal to 1.5x, patient is ineligible
  * ALK PHOS is greater than 5x ULN and AST or ALT is greater than 1.5x but less than or equal to 5x, patient is ineligible
  * ALK PHOS is greater than 5x ULN and AST or ALT is greater than 5x ULN, patient is ineligible
* Patients with neuropathy < 1.
* Ability to understand and the willingness to sign a written informed consent document
* Women of childbearing potential must have a negative pregnancy test
* Men and women of childbearing potential must be willing to consent to using effective contraception while on treatment and for at least 3 months thereafter

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks prior to entering the study
* Patients undergoing therapy with other investigational agents.
* Previous treatment involving regimen utilizing any of the protocol chemotherapeutic agents
* Patients with known brain metastases
* History of allergy to platinum compounds or to antiemetics appropriate for administration in conjunction with protocol-directed chemotherapy. Patients with a history of severe hypersensitivity reaction to Taxotere or Oxaliplatin or other drugs formulated with polysorbate 80
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, or unstable angina pectoris, or cardiac arrhythmia
* Pregnant and nursing women
* HIV-positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2004-09; Primary Completion 2009-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Gitlitz, MD, Principal Investigator — University of Southern California
Locations (1):
- USC/Norris Comprehensive Cancer Center, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at USC/Los Angeles County General Hospital and the USC/Norris Cancer Hopital between March 2005 and October 2007.
Pre-assignment Details: The trial had no pre-assignment criteria. All subjects were given the same treatment.
Groups:
- Taxotere Followed by Oxaliplatin: On Day 1 of each day treatment cycle, patients receive Taxotere 60 mg/m2 as a 1-hour IV infusion, followed by the administration of oxaliplatin 100 mg/m2. Oxaliplatin will be administered IV over 2 hours at a rate of 10mg/m2/min. This treatment regimen will be repeated every 21 days.
Period: Overall Study
Arm/Group | Taxotere Followed by Oxaliplatin
Started | 12
Completed | 2
Not Completed | 10
Not completed — Death | 1
Not completed — Lack of Efficacy | 4
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 1
Not completed — Non-compliance | 2

BASELINE CHARACTERISTICS:
Arm/Group | Taxotere Followed by Oxaliplatin
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 6
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Tumor Response
Description: All eligible patients who received the first dose of Taxotere will be included in the analysis.
  Tumor Response will be categorized as: Complete Response (CR), Partial Response (PR), Stable Disease (SD), Progressive Disease (PD), Early Death from Malignant Disease.
  Per RECIST criteria, CR = disappearance of all target and nontarget lesions; PR = at least a 30% decrease in the sum of the largest diameter (LD) of target lesions taking as reference the baseline sum LD; SD = neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD taking as references the smallest sum LD since the treatment started; PD = at least a 20% increase in the sum of LD of target lesions taking as references the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: 6 months after the last subject enrolled has gone off study
Measure: Number; unit: Participants
Groups:
- Arm 1: Single arm study
Arm/Group | Arm 1
Number analyzed (Participants) | 12
Participants
  Complete Response | 0
  Partial Response | 1
  Stable Disease | 5
  Progressive Disease | 2
  Early Offstudy (refused further therapy) | 3
  Early Death (due to malignant disease) | 1

2. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: Safety evaluation according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 3.0.
Time Frame: At end of every cycle
Population: All participants who started treatment
Measure: Number; unit: Participants
Arm/Group | Taxotere Followed by Oxaliplatin
Number analyzed (Participants) | 12
Participants | 7

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time the subject received the initial Taxotere and Oxaliplatin infusion and continued throughout the study until 30 days afer the last dose.
Arm/Group | Taxotere Followed by Oxaliplatin
Serious Adverse Events (participants affected / at risk) | 7/12
Other Adverse Events (participants affected / at risk) | 11/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Taxotere Followed by Oxaliplatin (N=12)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 3 (3)
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 1 (1)
Death not associated with CTCAE term (Death NOS) (General disorders) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Fatigue (General disorders) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 1 (2)
Infection (documented clinically or microbiologically) (Infections and infestations) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Leukocytes (total WBC) (Investigations) | 2 (2)
Mood Alteration (Agitation) (Psychiatric disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Neutrophils/Granulocytes (ANC/AGC) (Investigations) | 1 (1)
Phosphate, serum-low (Hypophosphatemia) (Metabolism and nutrition disorders) | 1 (1)
Potassium, serum-low (Hypokalemia) (Metabolism and nutrition disorders) | 1 (1)
Neuropathy: cranial (CN VII motor-face; sensory-taste) (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Taxotere Followed by Oxaliplatin (N=12)
Constipation (Gastrointestinal disorders) | 4 (4)
Flushing (Vascular disorders) | 1 (1)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 8 (10)
Hemoglobin (Blood and lymphatic system disorders) | 9 (14)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 6 (6)
Taste alteration (dysgeusia) (Nervous system disorders) | 4 (4)
Pain (muscle) (Musculoskeletal and connective tissue disorders) | 2 (2)
Platelets (Investigations) | 1 (1)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Leukocytes (total WBC) (Investigations) | 3 (3)
Pain (cardiac/heart) (Cardiac disorders) | 1 (2)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 5 (6)
Pain (Head/headache) (Nervous system disorders) | 3 (3)
Neuropathy: Sensory (Nervous system disorders) | 2 (2)
Pain (Abdomen NOS) (Gastrointestinal disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 4 (4)
Hearing: patients without baseline audiogram and not enrolled in monitoring program (Ear and labyrinth disorders) | 1 (1)
Heartburn/Dyspepsia (Gastrointestinal disorders) | 1 (1)
Mood Alteration (Anxiety) (Psychiatric disorders) | 3 (3)
Fever (in the absence of neutropenia) (General disorders) | 2 (2)
Alkaline Phosphatase (Investigations) | 1 (1)
Mood alteration (Agitation) (Psychiatric disorders) | 1 (1)
Mood alteration (Depression) (Psychiatric disorders) | 2 (2)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 (1)
Supraventricular and nodal arrythmia (Sinus tachycardia) (Cardiac disorders) | 2 (2)
Pain (neck) (Musculoskeletal and connective tissue disorders) | 1 (1)
Neuropathy: motor (Nervous system disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3)
Ataxia (incoordination) (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 2 (3)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 2 (4)
INR (International Normalized Ratio of Prothrombin) (Investigations) | 2 (2)
PTT (Partial Thromboplastin Time) (Investigations) | 1 (1)
Calcium, serum-low (hypcalcemia) (Metabolism and nutrition disorders) | 1 (1)
Bicarbonate, serum-low (Metabolism and nutrition disorders) | 1 (1)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 1 (1)
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 2 (3)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 2 (3)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 1 (1)
Weight Loss (Investigations) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 3 (3)
Pain (middle ear) (Ear and labyrinth disorders) | 1 (1)
AST, SGOT (serum glutamic oxaloacetic transaminase) (Investigations) | 3 (3)
Nail changes (Skin and subcutaneous tissue disorders) | 2 (3)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils (Soft Tissue NOS) (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes